CLINICAL TRIAL: NCT02540525
Title: Transobturator Sling Compared With Single-incision Mini-sling for the Treatment of Stress Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Transobturator Sling Compared With Single-incision Mini-sling for the Treatment of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Emerson Oliveira, Phd, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-2009
Record Dates: First submitted 2014-02-22; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Injury Due to Sling-shot
Keywords: stress incontinence; transobturator sling; single-incision mini-sling
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single incision mini-sling (Experimental): Experimental group: surgery to treat stress urinary incontinence with the Ophira mini sling systemt®
  Interventions: Device: Ophira
- Transobturator sling (Active Comparator): Control group: surgery to treat stress urinary incontinence with the Unitape T Plus®.
  Interventions: Device: Transobturator sling

INTERVENTIONS:
Device: Ophira — The procedure will be perfomed with a single incision in anterior wall vagina
  Arms: Single incision mini-sling
Device: Transobturator sling — Safyre T Plus ® system uses two helical needles for securing an average urethral sling mesh polypropylene soft tissue below the pubic bone by means of spinal anesthesia. Short form of the sling implantation is carried out as follows: a small longitudinal incision in the anterior vaginal wall approximately 2 cm is performed at 1 cm from the urethral meatus. Takes place below minimum dissection toward the lower branch of the ischium, and with the aid of the needle obturator and perforated membrane (outside-in maneuver). After that, the sling is attached to the needle carrying the same path. Subsequently, the passage of the needle is held in contraleral side. The procedure finishes performing the adjustment of the track with the aid of Kelly forceps type.
  Other Names: Unitape T plus
  Arms: Transobturator sling

SUMMARY:
1. OBJECTIVE:

   To determine the efficacy and safety of a single-incision mini-sling compared with a transobturator midurethral sling for stress urinary incontinence (SUI) treatment.
2. METHODS:

This prospective single-center randomized controlled trial will involve 100 women with a diagnosis of SUI. Primary outcomes were the objective and subjective cure rates, defined as negative cough stress and pad tests, and satisfaction rates. Quality of life assessed by the Incontinence Quality of Life Questionnaire and the Urogenital Distress Inventory Short Form, operation time, complications, and reoperation rates were also recorded. The efficacy was analyzed using a noninferiority test with a margin of 15%. For the noninferiority test, a P value >.05 rejects the noninferiority hypothesis of the mini-sling.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Clinical and urodynamic diagnosis of stress urinary incontinence
* Absence of associated neurological diseases
* No clinically significant detrusor instability (ie, to determine which symptoms are proportionally more significant for patient incontinence efforts)

Exclusion Criteria:

* urodynamic changes suggesting a reduction in bladder capacity, bladder compliance or suggestive of bladder outlet obstruction
* Coagulopathies
* Pregnancy
* History of sensitivity to foreign body
* Acute Urinary Tract Infection
* Sequelae of high exposure to ionizing radiation
* Use of drugs that can result in high and / or risk of significant postoperative complications surgical risk, including any drug that interferes with blood clotting
* anesthetic contraindication to the procedure
* Vulvovaginitis: presence of vaginal discharge with laboratory proven infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the cure rates between the mini sling and classical transobturator tapes | Up to one year
  Percentage of patients who are regarded as cured or improved based on the following criteria:
  * Negative Cough Stress test 1 year after surgery
  * Pad Test < 2 g 1 year after surgery

SECONDARY OUTCOMES:
Number of participants with adverse events | 0, 1, 6 and 12 months after surgery
  Comparison of the intra- and postoperative complications between procedures

CONTACTS AND LOCATIONS:
Overall Officials: EMERSON OLIVEIRA, PhD, Principal Investigator — FACULTY OF MEDICINE OF ABC
Locations (1):
- Faculty of Medicine of ABC, Santo André, São Paulo, Brazil

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839